CLINICAL TRIAL: NCT00451906
Title: Open-label Study of Bevacizumab (AVASTIN®) in Combination With Platinum-containing Chemotherapy as First-line Treatment of Patients With Advanced or Recurrent Non-squamous Non-small Cell Lung Cancer
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Platinum-Containing Chemotherapy in Patients With Advanced or Recurrent Non-Squamous Cell Lung Cancer.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO19390
Record Dates: First submitted 2007-03-22; First posted 2007-03-26 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Platinum Compounds; Bevacizumab

ARMS (1):
- Bevacizumab + Chemotherapy (Experimental): Participants with advanced or recurrent NSCLC will be administered bevacizumab infusions at a dose of 7.5 milligram per kilogram (mg/kg) or 15 mg/kg (investigator's choice) on Day 1 and then every 3 weeks, intravenously (IV) for a maximum of 6 cycles in combination with the standard of care NSCLC first-line chemotherapy in line with the licensed national prescribing information, during the treatment period. The initial dose of bevacizumab will be administered following chemotherapy; all subsequent doses could be given before or after chemotherapy.
  Interventions: Drug: Platinum-based chemotherapy; Drug: Bevacizumab [Avastin]

INTERVENTIONS:
Drug: Platinum-based chemotherapy — As prescribed
Drug: Bevacizumab [Avastin] — 15 mg/kg IV on Day 1 of each 3 week cycle

SUMMARY:
This single arm study will assess the safety and efficacy of Avastin combined with platinum-containing chemotherapy regimens in patients with advanced or recurrent non-squamous non-small cell lung cancer (NSCLC). Avastin will be given as first-line treatment in combination with platinum-based chemotherapy or in combination with any standard of care NSCLC first-line chemotherapy used in line with the licensed national prescribing information. Eligible patients will receive Avastin (15mg/kg iv on day 1 of each 3 week cycle) concomitantly with chemotherapy. Avastin treatment will continue after completion of chemotherapy cycles until disease progression, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* histologically or cytologically documented inoperable, locally advanced ( stage III), metastatic (stage IV) or recurrent NSCLC other than squamous cell (tumors of mixed histology should be categorized by the predominant cell type);
* ECOG PS status 0-2;
* life expectancy >= 12weeks;
* adequate renal, liver and hematological function.

Exclusion Criteria:

* mixed, non-small and small cell tumors, or mixed adenosquamous carcinomas with a predominant squamous component;
* hemoptysis (>=1/2 teaspoon of bright red blood) in previous 3 months;
* evidence of tumor invading major blood vessels on imaging;
* evidence of CNS metastases, even if previously treated.
* major surgery (including open biopsy), significant traumatic injury within 28 days prior to enrolment, or anticipation of need for major surgery during study treatment;
* prior chemotherapy for stage IIIb/IV disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2252 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (305):
- Argentina (4):
  - Buenos Aires
  - Chaco-resistencia
  - Córdoba
  - San Miguel de Tucumán
- Australia (11):
  - St Leonards, New South Wales
  - Waratah, New South Wales
  - Auchenflower, Queensland
  - Chermside, Queensland
  - Tugun, Queensland
  - Box Hill, Victoria
  - Geelong, Victoria
  - Malvern, Victoria
  - Wodonga, Victoria
  - Perth, Western Australia
  - Sydney, New South Wales
- Austria (15):
  - Bludesch
  - Bregenz
  - Feldkirch
  - Graz
  - Innsbruck
  - Knittelfeld
  - Kufstein
  - Linz
  - Natters
  - Salzburg
  - Sankt Veit an der Glan
  - Vienna
  - Vöcklabruck
  - Wels
  - Zams
- Bosnia and Herzegovina (2):
  - Banja Luka
  - Sarajevo
- Brazil (14):
  - Fortaleza, Ceará
  - Vitória, Espírito Santo
  - Salvador, Bahia, Estado de Bahia
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Ijuí, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - Jaú, São Paulo
  - Ribeirão Preto, São Paulo
  - Santos, São Paulo
  - São Paulo, São Paulo
- Canada (2):
  - Vancouver, British Columbia
  - Montreal, Quebec
- China (4):
  - Beijing
  - Guangzhou
  - Hangzhou
  - Shanghai
- Colombia (3):
  - Bogotá
  - Cali
  - Manizales
- Czechia (3):
  - Brno
  - Pilsen
  - Prague
- Denmark (4):
  - Aarhus
  - Herlev
  - Hillerød
  - Næstved
- Ecuador (2):
  - Guayaquil
  - Quito
- Cairo, Egypt
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (4):
  - Helsinki
  - Paimio
  - Pori
  - Tampere
- France (27):
  - Aix-en-Provence
  - Avignon
  - Besançon
  - Béziers
  - Bordeaux
  - Brest
  - Caen
  - Chalon-sur-Saône
  - Clermont-Ferrand
  - Gap
  - Grenoble
  - Le Chesnay
  - Lille
  - Lyon
  - Marseille
  - Meaux
  - Nancy
  - Neuilly-sur-Seine
  - Paris
  - Perpignan
  - Reims
  - Saint-Julien-en-Genevois
  - Strasbourg
  - Toulon
  - Toulouse
  - Valenciennes
  - Vandœuvre-lès-Nancy
- Germany (42):
  - Augsburg
  - Bad Berka
  - Bayreuth
  - Berlin
  - Bielefeld
  - Bonn
  - Cologne
  - Coswig
  - Donaustauf
  - Düsseldorf
  - Ebensfeld
  - Erlangen
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Gauting
  - Gerlingen
  - Göttingen
  - Großhansdorf
  - Halle
  - Hamburg
  - Hanover
  - Karlsruhe
  - Kiel
  - Leer
  - Leipzig
  - Leverkusen
  - Löwenstein
  - Magdeburg
  - Mainz
  - Minden
  - München
  - Neuruppin
  - Nuremberg
  - Oldenburg
  - Rostock
  - Treuenbrietzen
  - Ulm
  - Villingen-Schwenningen
  - Wiesbaden
  - Wolfsburg
  - Würselen
- Hong Kong (2):
  - Hong Kong
  - Shatin
- Hungary (5):
  - Budapest
  - Mátraháza
  - Pécs
  - Szombathely
  - Törökbálint
- Reykjavik, Iceland
- Israel (7):
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Ramat Gan
  - Tel Aviv
  - Ẕerifin
- Italy (42):
  - Avezzano, Abruzzo
  - Pescara, Abruzzo
  - Bari, Apulia
  - Brindisi, Apulia
  - San Giovanni Rotondo, Apulia
  - Potenza, Basilicate
  - Rionero in Vulture, Basilicate
  - Catanzaro, Calabria
  - Avellino, Campania
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Carpi, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Rimini, Emilia-Romagna
  - Aviano, Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Sora, Lazio
  - Viterbo, Lazio
  - Genoa, Liguria
  - La Spezia, Liguria
  - Bergamo, Lombardy
  - Cremona, Lombardy
  - Milan, Lombardy
  - Pavia, Lombardy
  - S Fermo Della Battaglia, Lombardy
  - Sondrio, Lombardy
  - Novara, Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Catania, Sicily
  - Palermo, Sicily
  - Taormina, Sicily
  - Ancona, The Marches
  - Arezzo, Tuscany
  - Lido di Camaiore, Tuscany
  - Pisa, Tuscany
  - Camposampiero, Veneto
  - Feltre - Bl, Veneto
  - Negrar, Veneto
  - Bologna, Umbria
  - Forli, Emilia-Romagna
- Riga, Latvia
- Beirut, Lebanon
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Mexico (3):
  - Chihuahua City
  - León
  - Mexico City
- Netherlands (12):
  - Arnhem
  - Breda
  - Eindhoven
  - Groningen
  - Haarlem
  - Helmond
  - Hoofddorp
  - Nieuwegein
  - Schiedam
  - The Hague
  - Tiel
  - Zwolle
- Poland (6):
  - Bialystok
  - Krakow
  - Lublin
  - Poznan
  - Warsaw
  - Zabrze
- Portugal (7):
  - Braga
  - Coimbra
  - Lisbon
  - Porto
  - Santa Maria da Feira
  - Setúbal
  - Vila Nova de Gaia
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Timișoara
- Russia (12):
  - Balashikha
  - Engel's
  - Irkutsk
  - Kislino, Kursk Region
  - Krasnodar
  - Moscow
  - Samara
  - Smolensk
  - Stavropol
  - Tver'
  - Tyumen
  - Ulyanovsk
- Belgrade, Serbia
- Slovakia (4):
  - Bratislava
  - Košice
  - Nitra
  - Poprad
- Slovenia (2):
  - Golnik
  - Ljubljana
- Spain (22):
  - Alicante, Alicante
  - Elche, Alicante
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Manresa, Barcelona
  - Mataró, Barcelona
  - Sabadell, Barcelona
  - Terrassa, Barcelona
  - Santander, Cantabria
  - Girona, Girona
  - Huesca, Huesca
  - A Coruña, La Coruña
  - Lugo, Lugo
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Murcia, Murcia
  - Pamplona, Navarre
  - Salamanca, Salamanca
  - San Cristóbal de La Laguna, Tenerife
  - Valencia, Valencia
  - Barakaldo, Vizcaya
  - Zaragoza, Zaragoza
- Sweden (7):
  - Gothenburg
  - Lund
  - Malmo
  - Örebro
  - Stokholm, Solna
  - Umeå
  - Uppsala
- Switzerland (4):
  - Aarau
  - Baden
  - Genolier
  - Locarno
- Taiwan (4):
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (5):
  - Ankara
  - Gaziantep
  - Istanbul
  - Izmir
  - Sıhhiye, Ankara
- United Kingdom (8):
  - Aberdeen
  - Belfast
  - Birmingham
  - Cambridge
  - Cardiff
  - Manchester
  - Nottingham
  - Suffolk
- Venezuela (3):
  - Barcelona
  - Barquisimeto
  - Porlamar

REFERENCES:
- [Derived] Bearz A, Passalacqua R, Alabiso O, Cinieri S, Gridelli C, Cravesana C, Crino L. First-line bevacizumab-based therapy in advanced non-squamous non-small-cell lung cancer : analysis of the Italian patients enrolled in the SAiL study. Clin Drug Investig. 2012 Nov;32(11):755-60. doi: 10.1007/s40261-012-0001-9. PMID 23018280
- [Derived] Crino L, Dansin E, Garrido P, Griesinger F, Laskin J, Pavlakis N, Stroiakovski D, Thatcher N, Tsai CM, Wu YL, Zhou C. Safety and efficacy of first-line bevacizumab-based therapy in advanced non-squamous non-small-cell lung cancer (SAiL, MO19390): a phase 4 study. Lancet Oncol. 2010 Aug;11(8):733-40. doi: 10.1016/S1470-2045(10)70151-0. Epub 2010 Jul 23. PMID 20650686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 384 sites in 39 countries from 21 August 2006 to 30 June 2009.
Pre-assignment Details: A total of 2252 participants were enrolled into the study, of which 2172 received the study drug. A total of 80 randomized participants did not receive study drug.
Groups:
- Bevacizumab + Chemotherapy: Eligible participants with advanced or recurrent non-squamous non-small cell lung cancer (NSCLC) were administered bevacizumab infusions at a dose of 7.5 milligram per kilogram (mg/kg) or 15 mg/kg (investigator's choice) on Day 1 and then every 3 weeks, intravenously (IV) for a maximum of 6 cycles in combination with the standard of care NSCLC first-line chemotherapy in line with the licensed national prescribing information, during the treatment period. The initial dose of bevacizumab was to be administered following chemotherapy; all subsequent doses could be given before or after chemotherapy. After the end of chemotherapy participants without disease progression could continue bevacizumab as maintenance therapy until confirmed disease progression, unacceptable toxicity or participant consent withdrawal. Participants were followed-up through a final-visit (28 days after last bevacizumab infusion) and then every 3 months until death.
Period: Overall Study
Arm/Group | Bevacizumab + Chemotherapy
Started | 2252
Completed | 13
Not Completed | 2239
Not completed — Adverse Event | 515
Not completed — Lost to Follow-up | 31
Not completed — Withdrawal by Subject | 111
Not completed — Protocol Violation | 21
Not completed — Progressive disease | 1328
Not completed — Termination of the study | 108
Not completed — Other Reasons | 121
Not completed — Did not complete final visit | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were described for the intent-to-treat (ITT) population, which included all participants with at least one valid post-baseline (Day -28 to -1) assessment.
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 2172
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 866
  Male | 1306

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Special Interest
Description: Participants with adverse events (AEs) of special interest (hypertension, proteinuria, wound healing complications, gastrointestinal perforation, arterial and venous thromboembolic events, hemoptysis, Central Nervous System (CNS) bleeding, other hemorrhage events and congestive heart failure) were reported.
Time Frame: Up to 3 years
Population: The ITT population included all participants with at least one valid post-baseline (Day -28 to -1) assessment.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 2172
participants
  Hypertension | 687
  Proteinuria | 672
  Wound healing complication | 26
  Gastrointestinal perforation | 30
  Arterial/Venous thromboembolic events | 274
  Hemoptysis | 176
  CNS bleeding | 7
  Other hemorrhage events | 744
  Congestive heart failure | 17

2. Primary Outcome: Number of Participants With Serious Adverse Events Related to Bevacizumab
Description: Participants with serious adverse events (SAEs) related to bevacizumab were reported for the duration of the study.
Time Frame: Up to 3 years
Population: The ITT population included all participants with at least one valid post-baseline (Day -28 to -1) assessment.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 2172
participants | 283

3. Secondary Outcome: Duration of Overall Survival
Description: Overall survival time was defined as time between first bevacizumab administration and date of death, irrespective of the cause of death. Participants for whom no death was captured on the clinical database were censored at the most recent date they were known to be alive.
Time Frame: Up to 3 years
Population: The ITT population included all participants with at least one valid post-baseline (Day -28 to -1) assessment. Participants available at the time of assessment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 1258
Months | 14.6 [13.8 to 15.3]

4. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as time between first bevacizumab administration and date of first occurrence of progressive disease. Participants who had not progressed at the time of study completion (including participants who died before progressive disease) or who were lost to follow-up were censored at the last bevacizumab administration date. Progressive disease is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Time to disease progression was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0.
Time Frame: Up to 3 years
Population: The ITT population was considered for analysis, which included all participants with at least one valid post-baseline (Day -28 to -1) assessment. Participants available at the time of assessment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 1501
Months | 7.8 [7.5 to 8.1]

5. Secondary Outcome: Number of Participants With Central Nervous System Bleeding
Description: The incidence of central nervous system (CNS) bleeding was reported for participants who developed CNS metastases during the study period and who did not have Computed Tomography (CT) or magnetic resonance imaging (MRI) techniques of the head performed at baseline.
Time Frame: Up to 3 years
Population: The ITT population was used for analysis, which included all participants with at least one valid post-baseline (Day -28 to -1) assessment. n = number of participants available at the time of assessment who were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 367
participants
  With CNS metastases (n = 281) | 12
  Without CT/MRI scans (n = 367) | 16

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: The ITT population was used for the safety analysis, which included all participants who had been treated with bevacizumab and chemotherapy at least once.
Arm/Group | Bevacizumab + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 834/2212
Other Adverse Events (participants affected / at risk) | 1982/2212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=2212)
Anaemia (Blood and lymphatic system disorders) | 36
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 52
Leukopenia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 84
Pancytopenia (Blood and lymphatic system disorders) | 11
Thrombocythaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 44
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 8
Atrial flutter (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Cardiac failure congestive (Cardiac disorders) | 4
Cardiac flutter (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 3
Cardiogenic shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 17
Myocardial ischaemia (Cardiac disorders) | 4
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Tympanic membrane disorder (Ear and labyrinth disorders) | 1
Angle closure glaucoma (Eye disorders) | 1
Optic ischaemic neuropathy (Eye disorders) | 1
Retinal vein thrombosis (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Visual disturbance (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 3
Anal fistula (Gastrointestinal disorders) | 1
Anal stenosis (Gastrointestinal disorders) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Appendicitis perforated (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 3
Colitis ischaemic (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 18
Diverticular perforation (Gastrointestinal disorders) | 3
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8
Gastrointestinal perforation (Gastrointestinal disorders) | 9
Gingival disorder (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 4
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 2
Jejunal perforation (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 7
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 25
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 7
Small intestinal perforation (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 26
Aplasia (General disorders) | 1
Asthenia (General disorders) | 2
Catheter thrombosis (General disorders) | 4
Chest pain (General disorders) | 19
Chills (General disorders) | 1
Cyst rupture (General disorders) | 1
Death (General disorders) | 14
Extravasation (General disorders) | 1
Fatigue (General disorders) | 19
Feeling abnormal (General disorders) | 1
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 13
Hyperpyrexia (General disorders) | 1
Ill-defined disorder (General disorders) | 2
Impaired healing (General disorders) | 1
Infusion related reaction (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Multi-organ failure (General disorders) | 1
Pain (General disorders) | 3
Performance status decreased (General disorders) | 2
Pyrexia (General disorders) | 37
Sudden death (General disorders) | 4
Alcoholic liver disease (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 3
Hepatic failure (Hepatobiliary disorders) | 2
Hepatitis acute (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Abscess (Infections and infestations) | 3
Abscess bacterial (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 4
Anal infection (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 2
Candidiasis (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 2
Catheter site infection (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Central line infection (Infections and infestations) | 3
Clostridial infection (Infections and infestations) | 2
Device related infection (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 2
Empyema (Infections and infestations) | 6
Enterocolitis infectious (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 6
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 7
Lobar pneumonia (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Lung abscess (Infections and infestations) | 1
Lung infection (Infections and infestations) | 5
Mumps (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Neutropenic infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 2
Penile abscess (Infections and infestations) | 1
Peridiverticular abscess (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 52
Pneumonia necrotising (Infections and infestations) | 1
Pneumonia primary atypical (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Pyopneumothorax (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 10
Sepsis (Infections and infestations) | 8
Septic shock (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Superinfection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Urosepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Viral skin infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Bone fissure (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Aspiration bronchial (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 9
Blood potassium decreased (Investigations) | 1
C-reactive protein increased (Investigations) | 3
Creatinine renal clearance decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haematology test abnormal (Investigations) | 1
Haemoglobin decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 11
Transaminases abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 4
Cachexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 9
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 5
Hypercreatininaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Starvation (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Fistula (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphonia (Nervous system disorders) | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 4
Cerebral ischaemia (Nervous system disorders) | 4
Cerebral microangiopathy (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 7
Coma (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 8
Hemiparesis (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Hypertensive encephalopathy (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 2
Nervous system disorder (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 11
Toxic encephalopathy (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 7
Emotional disorder (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephritic syndrome (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Nephrotic syndrome (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 11
Renal failure acute (Renal and urinary disorders) | 8
Renal haemorrhage (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 18
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 4
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 12
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 55
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Astringent therapy (Surgical and medical procedures) | 1
Catheter placement (Surgical and medical procedures) | 1
Knee operation (Surgical and medical procedures) | 1
Lung lobectomy (Surgical and medical procedures) | 1
Pleurodesis (Surgical and medical procedures) | 1
Tumour excision (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 1
Capillary leak syndrome (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 29
Embolism (Vascular disorders) | 3
Embolism venous (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 2
Hypertension (Vascular disorders) | 9
Hypertensive crisis (Vascular disorders) | 4
Infarction (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 2
Peripheral vascular disorder (Vascular disorders) | 1
Phlebitis superficial (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 7
Vena cava thrombosis (Vascular disorders) | 1
Venous insufficiency (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 3
Venous thrombosis limb (Vascular disorders) | 2
Not Codable (Infections and infestations) | 1 — Neutropenia Due to Respiratory Infection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=2212)
Constipation (Gastrointestinal disorders) | 423
Diarrhoea (Gastrointestinal disorders) | 347
Nausea (Gastrointestinal disorders) | 827
Stomatitis (Gastrointestinal disorders) | 260
Vomiting (Gastrointestinal disorders) | 516
Chest pain (General disorders) | 224
Fatigue (General disorders) | 893
Pyrexia (General disorders) | 263
Alanine aminotransferase increased (Investigations) | 159
Aspartate aminotransferase increased (Investigations) | 141
Blood creatinine increased (Investigations) | 186
Gamma-glutamyltransferase increased (Investigations) | 121
Haemoglobin decreased (Investigations) | 788
Neutrophil count decreased (Investigations) | 696
Platelet count decreased (Investigations) | 573
Protein urine present (Investigations) | 111
White blood cell count decreased (Investigations) | 623
Anorexia (Metabolism and nutrition disorders) | 462
Hyperglycaemia (Metabolism and nutrition disorders) | 122
Arthralgia (Musculoskeletal and connective tissue disorders) | 182
Back pain (Musculoskeletal and connective tissue disorders) | 219
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 134
Myalgia (Musculoskeletal and connective tissue disorders) | 135
Pain in extremity (Musculoskeletal and connective tissue disorders) | 189
Dizziness (Nervous system disorders) | 128
Headache (Nervous system disorders) | 309
Neuropathy (Nervous system disorders) | 179
Insomnia (Psychiatric disorders) | 112
Proteinuria (Renal and urinary disorders) | 568
Cough (Respiratory, thoracic and mediastinal disorders) | 328
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 130
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 279
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 589
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 167
Alopecia (Skin and subcutaneous tissue disorders) | 526
Rash (Skin and subcutaneous tissue disorders) | 167
Hypertension (Vascular disorders) | 680

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.